CLINICAL TRIAL: NCT02799433
Title: Evaluation of the Healthy Apple Program to Improve Nutrition and Physical Activity Practices and Child Weight Change in Child Care Centers in San Francisco
Brief Title: Evaluation of the Healthy Apple Program in San Francisco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Jodi Stookey, Senior Epidemiologist, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTG HAP20112015
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Childhood Obesity
Keywords: Water; Physical activity; Child care; Weight change
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Body Weight Changes | interventions — retinoic acid receptor beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Services (Active Comparator): This group of child care centers receives standard services from the San Francisco Department of Public Health Child Care Health Program. CCHP offers services to child care centers annually. The standard services include nurse consultation, health education, monitoring of nutrition and physical activity resource need, vision, hearing, oral health, and height and weight screenings.
  Interventions: Behavioral: Usual services
- Usual services + HAP (Experimental): This group of child care centers receives all the standard services plus invitation to participate in the voluntary Healthy Apple Program (HAP). The Healthy Apple program involves child care provider self-assessment, followed by an iterative process of goal setting, technical assistance/training, and re-assessment.
  Interventions: Behavioral: Usual services + HAP

INTERVENTIONS:
Behavioral: Usual services + HAP — The HAP process includes child care center providers completing a self-assessment(s), setting improvement goals, receiving technical assistance materials, attending topic-specific workshops, improving best practices, re-self-assessment and qualification for a HAP award.
  Arms: Usual services + HAP
Behavioral: Usual services — Control condition
  Arms: Usual Services

SUMMARY:
This randomized controlled trial uses administrative public health screening data to test whether the Healthy Apple program (HAP), designed to support local implementation of national Let's Move! Child Care guidelines in San Francisco (SF), improves child care center nutrition and physical activity practices and child weight change.

DETAILED DESCRIPTION:
In the USA, First Lady Michelle Obama started a nationwide child care initiative called 'Let's Move! Child Care' which aims to improve nutrition and physical activity practices in child care centers to promote healthy weight for children ages 0-5y.

The San Francisco Child Care Wellness Collaborative, including the San Francisco Department of Public Health (SFDPH) and SF Children's Council, developed a citywide Healthy Apple Program (HAP) to support local implementation of the Let's Move! initiative.

The San Francisco Department of Public Health (SFDH) has an existing Child Care Health Program (CCHP) which provides nurse consultation and health education materials for child care centers and annual health screenings for children.

The aim of this analysis is to see whether child care centers offered the HAP in addition to usual CCHP services can improve child care center nutrition and physical activity practices and child weight change better than usual CCHP services alone.

ELIGIBILITY:
Inclusion Criteria:

* Child care center received nutrition screening services from the SFDPH Child Care Health Program in 2011-2012.

Exclusion Criteria:

* Child care center declines CCHP services in 2012-2015.
* Child care center is ineligible for CCHP services (based on funding source)
* Child care center is closed or not serving children
* Child or family decline the voluntary services

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3493 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
BMI percentile change | Fall to Spring (about 6 months)
  Annually, child BMI percentile is measured in Fall and about 6 months later in Spring.

SECONDARY OUTCOMES:
Incident overweight or obesity | 6 months
  New cases of overweight or obesity that developed between the Fall and Spring screening during the school year. % of children who are normal weight in Fall who become overweight or obese by Spring.

OTHER OUTCOMES:
Number of best practices | 6 months
  Child care center best practices, including use of physical activity curricula or pitchers of drinking water, and staff practice of joining in active play with children.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Stookey, PhD, Principal Investigator — San Francisco Department of Public Health
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
The data used for this analysis are public health program screening data.

REFERENCES:
- [Background] Ammerman AS, Ward DS, Benjamin SE, Ball SC, Sommers JK, Molloy M, Dodds JM. An intervention to promote healthy weight: Nutrition and Physical Activity Self-Assessment for Child Care (NAP SACC) theory and design. Prev Chronic Dis. 2007 Jul;4(3):A67. Epub 2007 Jun 15. PMID 17572971
- [Background] Alkon A, Crowley AA, Neelon SE, Hill S, Pan Y, Nguyen V, Rose R, Savage E, Forestieri N, Shipman L, Kotch JB. Nutrition and physical activity randomized control trial in child care centers improves knowledge, policies, and children's body mass index. BMC Public Health. 2014 Mar 1;14:215. doi: 10.1186/1471-2458-14-215. PMID 24580983
- See also: Website for the Let's Move! Child Care initiative — https://healthykidshealthyfuture.org/